CLINICAL TRIAL: NCT04210388
Title: A Randomized, Single-dose, Open-label, Single-center, Crossover Study to Assess the Relative Bioavailability and Safety of Different Formulations of AZD5718 in Healthy Volunteers
Brief Title: A Study to Assess the Amount of Drug Levels in Blood and Safety of AZD5718 Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D7550C00008
Record Dates: First submitted 2019-12-23; First posted 2019-12-24 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Relative Bioavailability; Crossover Study; Safety
MeSH Terms: conditions — Coronary Artery Disease | interventions — AZD5718

STUDY DESIGN:
Intervention Model Description: The overall treatment period will start with a 2-period, 2-dose treatment crossover, followed by a 3-period, 3-dose treatment crossover.
  The following treatments will be given:
  Treatment A: AZD5718 (Formulation A) Treatment B: AZD5718 (Formulation B) Treatment C: AZD5718 (Formulation C) Treatment D: AZD5718 (Formulation D) AZD5718 (AZD5718 film-coated tablet, Reference treatment)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AZD5718 tablet, Treatment A (Experimental): Volunteers will receive single doses of AZD5718 tablet, Formulation A under fasted conditions.
  Interventions: Drug: AZD5718 tablet, Formulation A
- AZD5718 tablet, Treatment B (Experimental): Volunteers will receive single doses of AZD5718 tablet, Formulation B under fasted conditions.
  Interventions: Drug: AZD5718 tablet, Formulation B
- AZD5718 tablet, Treatment C (Experimental): Volunteers will receive single doses of AZD5718 tablet, Formulation C under fasted conditions.
  Interventions: Drug: AZD5718 tablet, Formulation C
- AZD5718 tablet, Treatment D (Experimental): Volunteers will receive single doses of AZD5718 tablet, Formulation C under fasted conditions.
  Interventions: Drug: AZD5718 tablet, Formulation D
- AZD5718 film-coated tablet (Active Comparator): Volunteers will receive single doses of AZD5718 film-coated tablet, Reference treatment under fasted conditions.
  Interventions: Drug: AZD5718 film-coated tablet, Reference treatment

INTERVENTIONS:
Drug: AZD5718 tablet, Formulation A — Volunteers will receive single doses of AZD5718 tablet, Formulation A under fasted conditions. The dose will be administered with 240 mL (8 fluid ounces) of non-carbonated water after an overnight fast of at least 10 hours.
  Arms: AZD5718 tablet, Treatment A
Drug: AZD5718 tablet, Formulation B — Volunteers will receive single doses of AZD5718 tablet, Formulation B under fasted conditions. The dose will be administered with 240 mL (8 fluid ounces) of non-carbonated water after an overnight fast of at least 10 hours.
  Arms: AZD5718 tablet, Treatment B
Drug: AZD5718 tablet, Formulation C — Volunteers will receive single doses of AZD5718 tablet, Formulation C under fasted conditions. The dose will be administered with 240 mL (8 fluid ounces) of non-carbonated water after an overnight fast of at least 10 hours.
  Arms: AZD5718 tablet, Treatment C
Drug: AZD5718 tablet, Formulation D — Volunteers will receive single doses of AZD5718 tablet, Formulation D under fasted conditions. The dose will be administered with 240 mL (8 fluid ounces) of non-carbonated water after an overnight fast of at least 10 hours.
  Arms: AZD5718 tablet, Treatment D
Drug: AZD5718 film-coated tablet, Reference treatment — Volunteers will receive single doses of AZD5718 film-coated tablet, Reference treatment under fasted conditions. The dose will be administered with 240 mL (8 fluid ounces) of non-carbonated water after an overnight fast of at least 10 hours.
  Arms: AZD5718 film-coated tablet

SUMMARY:
The study is a randomized, single-dose, open-label, combined 2x2 dose and 3x3 dose crossover design in fixed sequence. In this study, the relative bioavailability of different formulations of AZD5718 will be assessed in healthy volunteers in order to compare the exposure of Formulations A to D to the AZD5718 film-coated tablet formulation. The overall treatment period will start with a 2-period, 2-dose treatment crossover, followed by a 3-period, 3-dose treatment crossover.

DETAILED DESCRIPTION:
This study will be conducted at a single study center in Parexel Early Phase Clinical Unit London.

A total of 12 healthy male and female volunteers (of non-childbearing potential) will be randomized.

The study will comprise:

* A screening period of maximum 28 days
* Five treatment periods
* There will be a washout period of 3 to 6 days between dose administrations
* Follow-up visit, 5 to 7 days after last dose

Each volunteer will be involved in the study for between 7 and 9 weeks. The volunteers will be admitted to the Unit on the day before first dosing in Treatment Period 1 until at least 72 hours after last dosing in Treatment Period 5.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study volunteers should fulfill the following criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male or female volunteers aged 18 to 55 years (inclusive at screening) with suitable veins for cannulation or repeated venipuncture.
* Males must be willing to use appropriate contraception methods.
* Females must have a negative pregnancy test at screening and on admission to the Clinical Unit (Day -1), must not be lactating and must be of non childbearing potential, confirmed at screening by fulfilling the criteria.
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

Volunteers will not enter the study if any of the following exclusion criteria are fulfilled:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first dosing.
* Any clinically significant abnormalities in hematology, clinical chemistry, or urinalysis results, at screening or on admission to the Clinical Unit (Day -1), as judged by the Investigator, including:

  1. Alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN).
  2. Aspartate aminotransferase (AST) >1.5 x ULN.
  3. Total bilirubin (TBL) >1.5 x ULN.
  4. Gamma glutamyl transpeptidase (GGT) >1.5 x ULN. Out-of-range test may be repeated once for each visit at the discretion of the Investigator.
* Known or suspected Gilbert's syndrome.
* Any clinically significant abnormal findings in vital signs at screening or on admission to the Clinical Unit, as judged by the Investigator.
* Any clinically significant abnormalities on 12-lead ECG at screening, as judged by the Investigator.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
* Known or suspected history of drug abuse, as judged by the Investigator.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of first dosing in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5718.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the 3 months prior to screening.
* Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate) as judged by the Investigator.
* Positive screen for drugs of abuse or cotinine at screening or admission to the Clinical Unit or positive screen for alcohol on admission to the Clinical Unit.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to first dosing.
* Use of any prescribed or non prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to first dosing or longer if the medication has a long half-life.
* Known or suspected history of alcohol or excessive alcohol intake, as judged by the Investigator.
* Involvement of any AstraZeneca, Parexel or study site employee or their close relatives.
* Volunteers who have previously received AZD5718.
* Judgement by the Investigator that the volunteers should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Vulnerable volunteers, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from zero to infinity (AUC) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Area under the plasma concentration-curve from time zero to time of last quantifiable concentration (AUClast) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Maximum observed plasma concentration (Cmax) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Drug concentration at 24 hours after dosing (C24) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Time to reach maximum observed plasma concentration (tmax) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Terminal elimination rate constant (λz) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Dose normalized AUC (AUC/D) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Dose normalized AUClast (AUClast/D) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Dose normalized Cmax (Cmax/D) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers
Dose normalized C24 (C24/D) | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hours post-dose
  To evaluate the relative bioavailability of different formulations of AZD5718 and compare with the formulation used in the ongoing Phase 2a clinical study (Reference treatment), in healthy volunteers

SECONDARY OUTCOMES:
Number of volunteers with having adverse events and/or abnormal findings in vital signs and/or clinical laboratory assessments and/or physical examination and/or electrocardiogram (ECG) evaluation and/or body weight | From Screening up to 9 weeks
  To further assess the safety and tolerability of single doses of AZD5718 in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pablo Forte Soto, Principal Investigator — Senior Clinical Research Physician, Parexel Early Phase Clinical Unit London
Locations (1):
- Research Site, Harrow, United Kingdom